CLINICAL TRIAL: NCT00605930
Title: Energy Metabolism in Neurodegenerative Diseases: A Randomized, Double Blind, Placebo-Controlled Clinical Pilot Trial of Pyruvate, Creatine, and Niacinamide in Progressive Supranuclear Palsy.
Brief Title: A Pilot Clinical Trial of Pyruvate, Creatine, and Niacinamide in Progressive Supranuclear Palsy.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Louisville (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 083.03; 420
Record Dates: First submitted 2008-01-14; First posted 2008-01-31 (Estimated); Last update posted 2017-04-10 (Actual); Status verified 2017-04

CONDITIONS: Progressive Supranuclear Palsy
Keywords: Progressive Supranuclear Palsy; PSP; Nutriceutical; Pyruvate; Creatine; Niacinamide
MeSH Terms: conditions — Supranuclear Palsy, Progressive | interventions — Pyruvic Acid; Creatine; Niacinamide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Pyruvate, creatine, niacinamide (Active Comparator): Pyruvate, creatine, niacinamide administered
  Interventions: Dietary Supplement: Pyruvate, creatine, niacinamide
- Placebo (Placebo Comparator): placebo
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Pyruvate, creatine, niacinamide — A bar of 2 gm of pyruvate and 1 gm of creatine, and a pill of 1 gm of niacinamide once a day for 24 weeks.
  Arms: Pyruvate, creatine, niacinamide
Dietary Supplement: Placebo — 25% of subjects will receive a placebo bar and a placebo pill once a day for 24 weeks.
  Arms: Placebo

SUMMARY:
This study intends to study the safety and tolerance of the combination of pyruvate, creatine, and niacinamide over 6 months in patients with PSP.

DETAILED DESCRIPTION:
There are no effective symptomatic or biologic treatments for progressive supranuclear palsy (PSP), a relatively rare neurodegenerative disease that presents late in life with relentless progressive postural balance disturbances, non-levodopa responsive parkinsonism, supranuclear vertical gaze palsy, pseudobulbar palsy, and frontal behavioral and dysexecutive symptoms. In light of currently proposed etiopathogenic mechanisms in PSP and based on successful experiments inhibiting cellular neurotoxicity, it is hypothesized that preservation of brain energy homeostasis may allow endogenous neuroprotective mechanisms to reverse or impede free radical injury or other neurotoxic events leading to neurodegeneration in this disease. An emerging literature has described the neuroprotective effects of pyruvate, (as a neuronal energy fuel and free radical scavenger); niacinamide, (which boosts cofactor NAD), and creatine, (which buffers and selectively parcels cellular energy utilization) in various animal models of brain injury or degeneration.

Ajay Verma et al. have further demonstrated a synergistic neuroprotective effect of these three nutrients in various neural injury models. We thus propose using these nutrients as a novel and safe neuroprotective approach for treating PSP patients. This randomized, double-blind, placebo, control pilot study will test the safety and tolerance of this nutrient combination over 6 months in patients with PSP, and will measure their transport across the blood brain barrier. In addition to clinical and neuropsychological outcome measures, brain creatine will also be evaluated using magnetic resonance spectroscopy before and after therapy

ELIGIBILITY:
Inclusion Criteria:

* All subjects must meet the clinically definite or probable NINDS-SPSP PSP diagnostic research criteria that includes the presence of postural instability at disease onset, as well as supranuclear vertical ophthalmoparesis.
* All subjects must be able to tolerate oral feedings and be ambulatory
* All subjects or their caregivers must be able to read and understand the consent

Exclusion Criteria:

* Any contraindications to the use of pyruvate, creatine, and niacinamide
* the presence of a medical condition that can reasonably be expected to subject the patient to unwarranted risk or require frequent changes in medication.
* Pregnancy, nursing, or lack of effective contraception, if still at child-bearing age.
* History of prior sever traumatic brain injury or other severe neurologic or psychiatric condition, such as psychosis, stroke, multiple sclerosis, or spinal cord injury, which will interfere with outcome evaluation, in the opinion of the local principal investigator
* Subject unable to discontinue prohibited medication, which includes antiparkinsonian medications with potential neuroprotective effects such as amantadine, deprenyl, and vitamin E supplements > 400 IU per day.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2004-04; Primary Completion 2009-12 (Actual); Study Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
Clinical features of PSP, including motor function, neuropsychological function, and blood chemistry | Baseline, 4 weeks, 24 weeks

SECONDARY OUTCOMES:
CSF metabolite concentrations | Baseline, 24 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Irene Litvan, MD, Principal Investigator — University of Louisville, Division of Movement Disorders
Locations (1):
- Frazier Rehab, Louisville, Kentucky, United States

REFERENCES:
- See also: Related Info — http://www.litvanfoundation.com